CLINICAL TRIAL: NCT05826535
Title: A Phase 1/2 Multi-Center Study Evaluating the Safety and Efficacy of LYL314, a CD19/CD20 Dual-Targeting Chimeric Antigen Receptor T-Cell Therapy in Participants With Aggressive B-Cell Non-Hodgkin Lymphoma
Brief Title: Study of LYL314 in Aggressive Large B-Cell Lymphoma
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Lyell Immunopharma, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: LYL314-101
Record Dates: First submitted 2023-03-24; First posted 2023-04-24 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2025-11

CONDITIONS: Relapsed Non-Hodgkin Lymphoma; Refractory Non-Hodgkin Lymphoma; Non-Hodgkin Lymphoma; Large B-cell Lymphoma
Keywords: CAR T-cell; Non-Hodgkin Lymphoma; CD19/20; CD19; CD20; NHL; Diffuse Large B-cell lymphoma; DLBCL; Transformed follicular lymphoma; TFL; Primary mediastinal B-cell lymphoma; PMBCL; High-grade B-cell lymphoma; HGBL; follicular lymphoma Grade 3B; large cell follicular lymphoma; Aggressive B-cell NHL; Refractory Aggressive B-Cell Lymphoma; Refractory B-Cell Non-Hodgkin Lymphoma; Lymphoma, Non-Hodgkin; Lymphoma; Lymphoma, Large B-Cell, Diffuse; Cyclophosphamide; Fludarabine; Lymphoma, Follicular; Lymphoma, B-cell; Immunosuppressive Agents; Immunologic Factors; Disease Attributes; Immune System Diseases; Recurrence; PiNACLE
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Follicular; Lymphoma, B-Cell; Lymphoma; Disease Attributes; Immune System Diseases; Recurrence | interventions — fludarabine; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Phase 1 CAR T naïve (Cohort 1) (Experimental)
  Interventions: Drug: LYL314; Drug: Fludarabine; Drug: Cyclophosphamide
- Phase 1 CAR T experienced (Cohort 2) (Experimental)
  Interventions: Drug: LYL314; Drug: Fludarabine; Drug: Cyclophosphamide
- Phase 1 Refractory disease or relapse within one year of first-line therapy (Cohort 3) (Experimental)
  Interventions: Drug: LYL314; Drug: Fludarabine; Drug: Cyclophosphamide
- Phase 1 Received T-cell engager (TCE) therapy (Cohort 4) (Experimental)
  Interventions: Drug: LYL314; Drug: Fludarabine; Drug: Cyclophosphamide
- Phase 1 Receiving first-line treatment for high-risk large B-cell lymphoma (Cohort 5) (Experimental)
  Interventions: Drug: LYL314; Drug: Fludarabine; Drug: Cyclophosphamide
- Phase 2 CAR T naïve (Cohort 1) (Experimental): Single dose determined during Phase 1.
  Interventions: Drug: LYL314; Drug: Fludarabine; Drug: Cyclophosphamide

INTERVENTIONS:
Drug: LYL314 — CAR T-cell therapy
Drug: Fludarabine — Conditioning chemotherapy
Drug: Cyclophosphamide — Conditioning chemotherapy

SUMMARY:
This is a Phase 1/2, multi-center, open-label study evaluating the safety and efficacy of LYL314, a dual-targeting chimeric antigen receptor (CAR) targeting cluster of differentiation (CD)19 and CD20 in participants with aggressive large B-cell lymphoma.

DETAILED DESCRIPTION:
This is a Phase 1/2, multi-center, open-label study evaluating the safety and efficacy of LYL314, a dual-targeting chimeric antigen receptor (CAR) targeting cluster of differentiation (CD)19 and CD20 in participants with aggressive large B-cell lymphoma.

Five cohorts of participants will be enrolled:

Cohort 1: Participants who have not received a prior CAR T-cell product (CAR T naïve) and have received at least two or more prior lines of treatment (third-line or later).

Cohort 2: Participants who have received a prior CAR T-cell product (CAR T experienced) and have received at least two or more prior lines of treatment including one CAR T-cell therapy.

Cohort 3: Participants with refractory disease or relapse within one year of first-line therapy (second-line).

Cohort 4: Participants who have received prior T-cell engager (TCE) therapy and have received at least two or more prior lines of treatment including one TCE therapy.

Cohort 5: Participants receiving first-line treatment for high-risk large B-cell lymphoma who remain with disease on positron emission tomography scanning (PET-positive) after 2 to 3 cycles of standard-of-care chemoimmunotherapy (high-risk first-line).

Up to approximately 150 participants (across all cohorts) will be enrolled in the dose finding Phase 1 part of the study.

The Phase 2 pivotal study (PiNACLE) will expand enrollment of Cohort 1 to approximately 120 participants to further evaluate the safety and efficacy of LYL314.

LYL314 treatment consists of a single administration of CAR transduced autologous T-cells administered intravenously after a conditioning chemotherapy regimen consisting of fludarabine and cyclophosphamide, administered over 3 days.

Individual participants will remain in the active post-treatment follow-up (PTFU) period for approximately 2 years. Participants will continue in long-term follow-up (LTFU) for 15 years from LYL314 treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years or older at time of informed consent
2. Willing and able to provide written informed consent
3. Histologically confirmed aggressive NHL, including the following types defined by the World Health Organization (WHO 2017):

   * DLBCL
   * DLBCL arising from follicular lymphoma (transformed FL, tFL)
   * Primary mediastinal (thymic) large B-cell lymphoma (PMBCL)
   * High-grade large B-cell lymphoma with or without MYC and BCL2 and/or BCL6 rearrangement (HGBL)
   * Grade 3B follicular lymphoma/Large cell follicular lymphoma (FL3B)
4. Received at least two prior lines of therapy for Cohorts 1, 2, and 4 and one prior line of therapy for Cohort 3. Prior therapy must have included:

   * Anti-CD20 monoclonal antibody, and
   * An anthracycline containing chemotherapy regimen
   * Participants with tFL must have received at least one of their prior lines of therapy after transformation to DLBCL

     4b. Cohort 5 (High-risk first-line) participants must have high-risk large B-cell lymphoma
5. Relapsed or refractory disease, defined by the following:

   * Disease progression after last regimen (including salvage therapy after autologous stem cell transplantation [ASCT]). In participants who have only received front-line therapy, progression should be ≤ 12 months of first-line therapy (applicable for Cohort 3)
   * In patients who received one line of therapy, refractory disease is defined as failure to achieve at least a PR after at least 4 cycles of therapy (applicable for Cohort 3)
   * In patients who received two or more lines of therapy (Cohorts 1, 2, and 4), refractory disease is defined as failure to achieve a CR to last line of therapy (including CAR T and/or salvage therapy).
6. At least 1 measurable lesion (per Lugano classification). Lesions that have been previously irradiated will be considered measurable only if progression has been documented following completion of radiation therapy
7. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1 or ECOG 0 to 2 (Cohort 5)
8. Absolute neutrophil count (ANC) ≥ 1000/uL
9. Platelet count ≥ 50,000/uL
10. Absolute lymphocyte count (ALC) ≥ 200/uL

Other protocol-defined criteria apply.

Exclusion Criteria:

1. History of malignancy other than non-melanoma skin cancer or carcinoma in situ (e.g., cervix, bladder, breast) unless disease-free for at least 3 years. Participants who have received therapy for a prior malignancy within the prior 3 years, e.g., in the adjuvant setting, are not excluded
2. Active central nervous system (CNS) involvement by malignancy on magnetic resonance imaging (MRI) or by lumbar puncture. Participants with prior evidence of brain metastasis treated at least 8 weeks prior to enrollment will not be excluded for participation if CNS disease is deemed stable at the time of study enrollment
3. History of cardiac lymphoma involvement or Epstein-Barr virus (EBV)+ lymphoma
4. Ongoing or impending oncologic emergency (e.g., tumor mass effect, tumor lysis syndrome, known vascular invasion)
5. Received the following therapies in the specified time frame prior to enrollment/leukapheresis

   1. Any systemic therapy within 2 weeks
   2. Any systemic inhibitory/stimulatory immune checkpoint molecule therapy within 3 half-lives prior to enrollment (e.g., ipilimumab, nivolumab, pembrolizumab, atezolizumab, OX40 agonists, 4-1BB agonists)
   3. Fludarabine within 12 weeks
   4. Alemtuzumab, bendamustine or antithymocyte globuline (ATG) within 6 months
   5. Any T cell engager/bispecific antibody therapy such as CD20/CD3 or CD19/CD3 bispecific antibodies within 4 weeks
   6. Any experimental therapy within 4 weeks or 5 half-lives (whichever is shorter)
6. Received radiation therapy within 3 weeks prior to enrollment/leukapheresis
7. Experiencing non-hematologic toxicities due to prior therapy. Exceptions include: stable and recovered to grade ≤ 1 or non-clinically significant toxicities such as (1) alopecia, (2) toxicities where Grade 2 is solely defined by participant receiving hormone replacement therapy for endocrinopathies resulting from previous checkpoint inhibitor therapy, (3) Grade 2 lymphopenia, and (4) hearing loss or Grade 2 neuropathy associated with prior treatment with taxanes or platinating agents
8. History of allogeneic stem cell or solid organ transplantation
9. Receipt of autologous stem cell transplantation within 6 weeks prior to enrollment/leukapheresis
10. History of prior genetically modified cell therapy other than a product targeting CD19 with an FMC63-based CAR (e.g., axicabtagene ciloleucel (axi-cel), tisagenlecleucel (tisa-cel), or lisocabtagene maraleucel (liso-cel). For all other CAR T cell therapy treatments, discussion with the Sponsor's Medical Monitor is required
11. Primary immunodeficiency
12. History of autoimmune disease (e.g., Crohn's disease, rheumatoid arthritis, systemic lupus) resulting in end organ injury or requiring systemic immunosuppression/systemic disease modifying agents within the last 2 years. Participants who have other autoimmune condition(s) considered to be associated with underlying malignancy may be enrolled in the study after discussion with and approval of the Medical Monitor.

Other protocol-defined criteria apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 270 (Estimated)
Dates: Start 2023-05-09 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2031-06-30 (Estimated)

PRIMARY OUTCOMES:
Phase 1: Evaluate the safety and tolerability of a single dose of LYL314 administered as a single agent | Baseline to Month 24
  Incidence of dose-limiting toxicities (DLTs) and other treatment-emergent adverse events (TEAEs)
Phase 2: Estimate the efficacy of LYL314, as measured by ORR | Baseline to Month 24
  ORR based on Independent Review Committee (IRC) assessment per Lugano criteria

SECONDARY OUTCOMES:
Phase 1: Evaluate the efficacy of LYL314 | Baseline to Month 24
  Overall response rate (ORR), Complete response rate (CRR), duration of response (DOR), duration of complete response (DOCR), progression free survival (PFS) based on Investigator assessment until a pivotal trial (Phase 2) portion is initiated at which time all scans will be reviewed by an IRC assessment (Cohort 1) per Lugano criteria
Phase 1: Evaluate the feasibility of treatment with LYL314 | Baseline to Month 24
  Proportion of enrolled participants who receive the target dose of LYL314
Phase 1: Evaluate the pharmacokinetics of LYL314 when administered as a single agent | Baseline to Month 24
  Maximum concentration (Cmax), area under the curve from time 0 to Day 28 (AUC0-28) and persistence of LYL314
Phase 2: Estimate the efficacy of LYL314 | Baseline to Month 24
  ORR based on Investigator assessment per Lugano criteria
Phase 2: Estimate the efficacy of LYL314 | Baseline to Month 24
  DOR based on IRC assessment and investigator assessment per Lugano criteria
Phase 2: Estimate the efficacy of LYL314 | Baseline to Month 24
  Time to response (TTR) based on IRC assessment and investigator assessment per Lugano criteria
Phase 2: Estimate the efficacy of LYL314 | Baseline to Month 24
  PFS based on IRC assessment and investigator assessment per Lugano criteria
Phase 2: Estimate the efficacy of LYL314 | Baseline to Month 72
  Overall Survival (OS)
Phase 2: Evaluate the safety and tolerability of a single dose of LYL314 administered as a single agent | Baseline to Month 24
  Incidence and severity of TEAEs
Phase 2: Evaluate the pharmacokinetics of LYL314 when administered as a single agent | Baseline to Month 24
  Maximum concentration (Cmax), area under the curve from time 0 to Day 28 (AUC0-28) and persistence of LYL314

CONTACTS AND LOCATIONS:
Locations (26):
- United States (26):
  - University of California-Irvine Medical Center, Irvine, California
  - Cedars-Sinai Medical Center, Los Angeles, California
  - University of California, Los Angeles (UCLA) Medical Center, Los Angeles, California
  - Scripps Clinic, San Diego, California
  - Colorado Blood Cancer Institute, Denver, Colorado
  - Augusta University Medical Center, Augusta, Georgia
  - Indiana Blood and Marrow Transplantation, Indianapolis, Indiana
  - University of Iowa, Iowa City, Iowa
  - University of Louisville Brown Cancer Center, Louisville, Kentucky
  - Louisiana State University Health Sciences Center, Shreveport, Louisiana
  - Corewell Health, Grand Rapids, Michigan
  - University of Nebraska Medical Center, Omaha, Nebraska
  - University of New Mexico Comprehensive Cancer Center, Albuquerque, New Mexico
  - Montefiore Medical Center, The Bronx, New York
  - University of Cincinnati (UC) Physicians Company, LLC, Cincinnati, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - Lehigh Valley Topper Cancer Center Institute, Allentown, Pennsylvania
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - West Penn Hospital, Pittsburgh, Pennsylvania
  - Baylor University Medical Center, Dallas, Texas
  - Texas Transplant Institute, San Antonio, Texas
  - Huntsman Cancer Institute, Salt Lake City, Utah
  - Intermountain Healthcare, Salt Lake City, Utah
  - Virginia Oncology Associates, Norfolk, Virginia
  - Virginia Commonwealth University-Massey Cancer Center, Richmond, Virginia
  - Medical College of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No